CLINICAL TRIAL: NCT03287232
Title: Prasterone (DHEA) for the Treatment of Hypoactive Sexual Desire Disorder (HSDD) - (Placebo-Controlled, Double Blind and Randomized Phase III Study of Intravaginal Prasterone)
Brief Title: Prasterone (DHEA) for the Treatment of Hypoactive Sexual Desire Disorder (HSDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-242
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Prasterone; DHEA; Menopause; Sexual Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Vaginal Insert
- Prasterone (Experimental)
  Interventions: Drug: Prasterone 6.5 mg (0.50%) Vaginal Insert

INTERVENTIONS:
Drug: Placebo Vaginal Insert — Daily administration of a placebo vaginal insert.
  Arms: Placebo
Drug: Prasterone 6.5 mg (0.50%) Vaginal Insert — Daily administration of a 6.5 mg (0.50%) prasterone vaginal insert.
  Arms: Prasterone

SUMMARY:
The primary objective is to confirm the efficacy of intravaginal prasterone (DHEA) on Hypoactive Sexual Desire Disorder (HSDD) in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria (main criteria):

* Postmenopausal women (hysterectomized or not).
* Women between 40 and 80 years of age.
* Being in a stable relationship with the opportunity for sexual activity or masturbation at least once a month during the last 6 months or longer (before screening visit) and during the following 8 months.
* Diagnosis of HSDD confirmed by a qualified clinician.
* Willing to participate in the study and sign an informed consent.

Exclusion Criteria (main criteria):

* Chronic or acute life stress or major life change that could have interfered and continues to interfere significantly with sexual activity.
* Taking drugs which could be responsible for HSDD.
* Severe medical condition which can explain the loss of sexual desire.
* The administration of any investigational drug within 30 days of screening visit.
* Clinically significant abnormal serum biochemistry, urinalysis or hematology.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Sexual desire | 28 weeks
  Change from Baseline in sexual desire evaluated by the FSFI desire domain (Questions 1 & 2).
Distress from low sexual desire | 28 weeks
  Change from Baseline in distress from low sexual desire evaluated by question 13 of FSDS-DAO.

SECONDARY OUTCOMES:
Satisfying sexual events (SSEs) | 28 weeks
  Change from Baseline in the number of SSEs from a daily log of sexual activity.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Labrie, M.D., Ph.D., Study Chair — EndoCeutics Inc.; Leonard R. Derogatis, Ph.D., Principal Investigator — Maryland Center for Sexual Health
Locations (69):
- United States (63):
  - Endoceutics site # 106, Huntsville, Alabama
  - Endoceutics site # 104, Mobile, Alabama
  - Endoceutics site # 117, Tucson, Arizona
  - Endoceutics site # 108, Berkeley, California
  - Endoceutics site # 121, Los Alamitos, California
  - Endoceutics site #128, Los Angeles, California
  - Endoceutics site # 30, San Diego, California
  - Endoceutics site # 17, San Diego, California
  - Endoceutics site # 36, Denver, Colorado
  - Endoceutics site # 52, Denver, Colorado
  - Endoceutics site # 125, New London, Connecticut
  - Endoceutics site # 7, Washington D.C., District of Columbia
  - Endoceutics site # 95, Bradenton, Florida
  - Endoceutics site # 120, Coral Gables, Florida
  - Endoceutics site # 99, Fort Myers, Florida
  - Endoceutics site # 26, Jacksonville, Florida
  - Endoceutics site # 60, Lake Worth, Florida
  - Endoceutics site #118, Miami Lakes, Florida
  - Endoceutics site # 54, North Miami, Florida
  - Endoceutics site # 92, Oviedo, Florida
  - Endoceutics site # 105, Sanford, Florida
  - Endoceutics site # 114, St. Petersburg, Florida
  - Endoceutics site # 89, West Palm Beach, Florida
  - Endoceutics site # 80, West Palm Beach, Florida
  - Endoceutics site # 90, West Palm Beach, Florida
  - Endoceutics site # 107, Decatur, Georgia
  - Endoceutics site # 119, Roswell, Georgia
  - Endoceutics site # 23, Sandy Springs, Georgia
  - Endoceutics site # 91, Savannah, Georgia
  - Endoceutics site # 111, Wichita, Kansas
  - Endoceutics site # 55, Wichita, Kansas
  - Endoceutics site # 88, Lexington, Kentucky
  - Endoceutics site # 86, Louisville, Kentucky
  - Endoceutics site # 103, Boston, Massachusetts
  - Endoceutics site # 22, Kalamazoo, Michigan
  - Endoceutics site # 123, Portsmouth, New Hampshire
  - Endoceutics site # 101, Berlin, New Jersey
  - Endoceutics site # 50, Neptune City, New Jersey
  - Endoceutics site # 44, New Brunswick, New Jersey
  - Endoceutics site # 81, Plainsboro, New Jersey
  - Endoceutics site # 20, New York, New York
  - Endoceutics site # 110, Poughkeepsie, New York
  - Endoceutics site # 97, Rochester, New York
  - Endoceutics site # 58, Raleigh, North Carolina
  - Endoceutics site # 115, Fargo, North Dakota
  - Endoceutics site # 116, Canton, Ohio
  - Endoceutics site # 100, Cleveland, Ohio
  - Endoceutics site # 5, Cleveland, Ohio
  - Endoceutics site # 93, Columbus, Ohio
  - Endoceutics site # 75, Philadelphia, Pennsylvania
  - Endoceutics site # 127, Bluffton, South Carolina
  - Endoceutics site # 126, Mt. Pleasant, South Carolina
  - Endoceutics site # 112, Myrtle Beach, South Carolina
  - Endoceutics site # 94, Chattanooga, Tennessee
  - Endoceutics site # 64, Jackson, Tennessee
  - Endoceutics site #124, Knoxville, Tennessee
  - Endoceutics site #122, Nashville, Tennessee
  - Endoceutics site # 82, Houston, Texas
  - Endoceutics site # 102, San Antonio, Texas
  - Endoceutics site # 96, Charlottesville, Virginia
  - Endoceutics site # 3, Norfolk, Virginia
  - Endoceutics site # 98, Norfolk, Virginia
  - Endoceutics site # 76, Seattle, Washington
- Canada (6):
  - Endoceutics site # 68, Sarnia, Ontario
  - Endoceutics site # 18, Lévis, Quebec
  - Endoceutics site # 02, Québec, Quebec
  - Endoceutics site # 77, Québec, Quebec
  - Endoceutics site # 78, Québec, Quebec
  - Endoceutics site # 11, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Effect of intravaginal dehydroepiandrosterone (Prasterone) on libido and sexual dysfunction in postmenopausal women. Menopause. 2009 Sep-Oct;16(5):923-31. doi: 10.1097/gme.0b013e31819e85c6. PMID 19424093
- [Background] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Background] Bouchard C, Labrie F, Derogatis L, Girard G, Ayotte N, Gallagher J, Cusan L, Archer DF, Portman D, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Group. Effect of intravaginal dehydroepiandrosterone (DHEA) on the female sexual function in postmenopausal women: ERC-230 open-label study. Horm Mol Biol Clin Investig. 2016 Mar;25(3):181-90. doi: 10.1515/hmbci-2015-0044. PMID 26725467